CLINICAL TRIAL: NCT06739551
Title: Comparison of Efficacy of Oral Methotrexate and Acitretin for Generalized Lichen Planus
Brief Title: Systemic Treatment Options for Generalized Lichen Planus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Mohibullah Zahidi, Post Graduate Resident in Dermatology, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SheikhZMC/H
Record Dates: First submitted 2024-12-05; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Lichen Planus
Keywords: Lichen Planus; Acitretin; Methotrexate; Efficacy
MeSH Terms: conditions — Lichen Planus | interventions — Methotrexate; Pharmaceutical Preparations; Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral methotrexate group (Group A) (Active Comparator): Patients with generalized lichen planus will be given 10 mg per week
  Interventions: Drug: Methotrexate (drug)
- Oral Acitretin group (Group B) (Active Comparator): Patients with generalized lichen planus will be given oral acitretin 50 mg once daily
  Interventions: Drug: Acitretin

INTERVENTIONS:
Drug: Methotrexate (drug) — oral methotrexate 10 mg per week for 12 weeks
  Arms: Oral methotrexate group (Group A)
Drug: Acitretin — oral acitretin 50 mg once daily for 12 weeks
  Arms: Oral Acitretin group (Group B)

SUMMARY:
Lichen planus is a chronic inflammatory skin condition with unknown etiology. It requires a long term treatment. Evaulating the most efficacious, safe and affordable treatment option is the need of the hour. This study is going to compare the efficacy of two familiar drugs (acitretin and methotrexate) in the treatment of generalized lichen planus as to find out the relatively more effective and safer treatment.

DETAILED DESCRIPTION:
Lichen planus (LP) is a chronic mucocutaneous condition of an unknown cause. It presents clinically as purple, itchy papules and plaques on the lower back, body folds, oral mucosa, and on the scalp(1). It is recurrent condition with a prolonged course and requires an effective, safer and relatively cheaper treatment option (2).

Objective: "To compare the efficacy of oral methotrexate vs. oral acitretin in the treatment of generalized lichen planus".

Material & Methods: This randomized comarative study will be carried out in Outpatient Dermatology Department, Sheikh Zayed Hospital Rahim Yar Khan, Pakistan. Approval of the study has been taken from ethical review committee of the hospital.Data will be collected on prescribed form. Patient will be selected on basis of inclusion & exclusion criteria. Informed consent will be taken from selected patients before data collection. Study will include 124 patients which will be divided into 2 groups A & B, 62 in each group. Group A will receive oral methotrexate 10mg once weekly for 12 weeks. Group B will receive oral acitretin 50mg daily for 12 weeks. Folic acid will be given to all patients in group A at a dose of five milligram per day. Patient will be followed at 4 weekly interval and final efficacy will be determined at 12th week.Data will be analyzed by SPSS v25.0.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years
* Gender: both male and female
* Type of Lichen planus: generalized lichen planus
* Patients not taking prior treatment in last 1 month

Exclusion Criteria:

* Pregnancy and lactating females
* Bleeding disorders
* Abnormal liver function tests
* Platelet count less than 100000
* Hypersensitivity to Methotrexate or Acitretin
* Unrealistic expectations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy of oral methotrexate vs. oral acitretin in the treatment of generalized lichen planus | Clinical assessment for efficacy will be done 4 weekly for 12 weeks.
  Efficacy will be assesssed clinically at each follow up visit. Final efficacy of each treatment will be determined at last follow up visit( i.e. at 12 th week after start of treatment).The final efficacy will be divided into following groups on the basis of clinical resolution of disease:
  1. Remission: It is defined as complete resolution of all lesions leaving behind normal skin or post inflammatory pigmentation.
  2. Improvement: It is defined as a more than 50% decrease of the disease, as clinically measured by the surface area from the baseline.
  3. No improvement: It is defined as less than a 50% improvement in the disease, as measured clinically by the surface area from the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh zayed Medical College and Hospital, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No